CLINICAL TRIAL: NCT07405177
Title: A Randomized, Open-label, Parallel-group Study to Assess the Pharmacokinetic Bioequivalence of Subcutaneously-administered Tulisokibart Delivered by 2 Different Autoinjectors in Healthy Participants
Brief Title: A Study of MK-7240 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7240-009; MK-7240-009 (Other: MSD)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Tulisokibart Form 1 (Experimental): Participants will receive tulisokibart form 1.
  Interventions: Biological: Tulisokibart Form 1
- Arm 2: Tulisokibart Form 2 (Experimental): Participants will receive tulisokibart form 2.
  Interventions: Biological: Tulisokibart Form 2

INTERVENTIONS:
Biological: Tulisokibart Form 1 — Solution for injection.
  Other Names: MK-7240
  Arms: Arm 1: Tulisokibart Form 1
Biological: Tulisokibart Form 2 — Solution for injection.
  Other Names: MK-7240
  Arms: Arm 2: Tulisokibart Form 2

SUMMARY:
The goal of this study is to learn what happens to MK-7240 in a healthy person's body over time (pharmacokinetic or PK study). Researchers also want to learn about the safety of MK-7240 and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Has a body-mass index (BMI) between 18 and 32 kg/m^2

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

* Has a history of more than 1 episode of herpes zoster infection or history of disseminated herpes zoster infection
* Has a history of or current active tuberculosis (TB) infection or history of latent TB that was not fully treated

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the AUC0-inf of tulisokibart.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the AUC0-last of tulisokibart.
Maximum Plasma Concentration (Cmax) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the Cmax of tulisokibart.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | At designated timepoints up to 14 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Due to an AE | At designated timepoints up to 14 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time to Maximum Plasma Concentration (Tmax) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the Tmax of tulisokibart.
Apparent Clearance (CL/F) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the CL/F of tulisokibart.
Apparent Volume of Distribution (V/F) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the V/F of tulisokibart.
Apparent Terminal Half-life (t1/2) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the t1/2 of tulisokibart.
Apparent Terminal Elimination Rate constant (Kel) of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the Kel of tulisokibart.
Ratio of AUC0-Last/AUC0-Inf of Tulisokibart | At designated timepoints up to 14 weeks
  Blood samples will be collected to determine the ratio of AUC0-last/AUC0-inf of tulisokibart.
Area Under the Concentration-Time Curve from Time 0 to Day 14 (pAUC0-14) of Tulisokibart | At designated timepoints up to 14 days
  Blood samples will be collected to determine pAUC0-14 of tulisokibart.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com